CLINICAL TRIAL: NCT02488278
Title: GLUCOME USABILITY STUDY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: GlucoMe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Clin-001-00
Record Dates: First submitted 2015-06-23; First posted 2015-07-02 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Glucose blood measurements, glucometers ,audio communication
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self-Monitoring of Glucose Blood Measurements (No Intervention): Self-Monitoring of Glucose Blood Measurements using the GlucoMe Glucose Monitoring Device and App
  Interventions: Device: GlucoMe Glucose Monitoring Device

INTERVENTIONS:
Device: GlucoMe Glucose Monitoring Device — Perform a blood glucose test using the application and device

SUMMARY:
The GlucoMe device, in its original packaging, along with the user manual and QuickStart guide will be provided to the patient in a simulated home use environment. The patient labeling will be in the format intended for distribution.

Ten (10) subjects identified as potential end users of the GlucoMe device will receive the user manual. An additional ten (10) subjects also identified as potential end users of the GlucoMe device will NOT receive the user manual. All subjects will be provided with a pre-test and post-test questionnaire and a list of tasks to complete, including applying and operating the device.

The observer and user post-test questionnaire will collect information regarding device use. The device's use will be compared with identified risks to determine if the percentage of failures is within the study protocol success criteria. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

DETAILED DESCRIPTION:
Twenty (20) subjects identified as potential end users of the device will be recruited to the study and screened according to the study inclusion and exclusion criteria. Subjects will be asked to sign informed consent. The GlucoMe device, in its original packaging, along with the user manual and QuickStart guide will be provided to the patient in a simulated home-use environment. The patient labeling will be in the format intended for distribution.

Ten (10) subjects identified as potential end users of the GlucoMe device will receive the user manual and QuickStart guide. An additional ten (10) subjects also identified as potential end users of the GlucoMe device will not receive the user manual, but will receive the QuickStart guide. All subjects will be provided with a pre-test and post-test questionnaire and a list of tasks to complete, including applying and operating the device.

The observer examination and user post-test questionnaire will collect information regarding device use. The device's use will be compared with identified risks to determine if the percentage of failures is within the study protocol success criteria. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female equal to or greater than 18 years of age.
2. Subject is a potential candidate for purchasing the GlucoMe device (e.g., subjects diagnosed with diabetes type 1 or 2).
3. Subject has facility with both hands.
4. Subject monitors himself.
5. Subject knows how to download and install apps.
6. Subject is capable of understanding and is willing to sign informed consent.

Exclusion Criteria:

1. Subject has dementia.
2. Subject has mental disorders.
3. Subject was diagnosed with diabetes other than type 1 or 2 (e.g. gestational diabetes, congenital diabetes, drug induced diabetes, etc.).
4. Subject does not monitor himself.
5. Subject is visually impaired.
6. Subject cannot draw blood samples from fingertip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Operating the GlucoMe device: obtaining a glucose reading and recording the results | 1 Hour
  Using the device, with or without the user manual, all 20 subjects tested were able to complete device related tasks, including starting the application, operating the GlucoMe device and obtaining a glucose reading and recording the results, in a timeframe of up to 1 hour and with minimal attempts to ask for assistance; and Using the device and the user manual. Considering that the GlucoMe is a low risk device, and the probability of an occurrence and the severity of a failure are low, a success rate of 100% potential end user subjects passing may be considered acceptable for the over the counter use of the device. Any failures to complete the device related tasks and/or self-exclude from use of the device must be explained.

SECONDARY OUTCOMES:
Time to completion of obtaining a glucose reading using the application and device | 1 Hour
  The following measurable usability criteria for specific, critical steps, based on observer evaluation or user post-test questionnaire responses, will be assessed through analysis of the data following the study:
  Time-to-completion of task; Time to completion of obtaining a glucose reading using the application and device will be measured by the observer for both arms and will be analysed
Frequency of attempts to ask for assistance during the use of the device and application | 1 hour
  Frequency of attempts to ask for assistance will be documented by the observer for both arms and will be analysed
Participants' level of success in completing tasks related to the use of the device and application | 1 hour
  Numerical ratings describing the participants' level of success in completing tasks will be collected through user post-test questionnaire responses, for both arms and will be analysed
Documenting specific user errors and inefficiencies related to the use of the device and application | 1 hour
  Qualitative information regarding specific user errors and inefficiencies will be collected through observer evaluation and user post-test questionnaire responses, for both arms and will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Ahava Stein, Study Director — A. Stein Regulatory Affairs Consulting Ltd.